CLINICAL TRIAL: NCT04901598
Title: Physical Activity Level, Aerobic Capacity and Dietary Habits Among a Cohort of Females With Premenstrual Syndrome: an Observational Study
Brief Title: Physical Activity Level, Aerobic Capacity and Dietary Habits Among a Cohort of Females With Premenstrual Syndrome
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nisreen Ashraf, principle investigator, Cairo University
Other Study IDs: p.t.REC/012/003220
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Premenstrual Syndrome
Keywords: physical activity level, aerobic capacity and dietary habits in PMS
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Running anaerobic sprint test and aerobic test — subjects walk a mile with maximum steps and their heart rate will not exceed 180 beats per minute during the test and the execution time will not be less than 9 minutes (RAST test)

SUMMARY:
The aim of the study is to investigate the physical activity level, aerobic capacity and dietary habits among a cohort of females with premenstrual syndrome

DETAILED DESCRIPTION:
premenstrual syndrome can be defined as a recurrent disorder that occurs every month in the luteal phase of the menstrual cycle, and subside with the onset of menstruation. It is characterized by a complex set of symptoms, which include physical, psychological and behavioral changes with varying severity. This can interfere with the lives of females. Physical exercise improves PMS through rising endorphin levels, reducing adrenal cortisol symptoms, leading to lesser anxiety, depression and greater pain tolerance, as previous studies showed that it was effective in decreasing pain as well as mental and physical symptoms of PMS. Recently, lifestyle changes have gained more importance than pharmacotherapy. Lifestyle changes include many methods including diet regulation and exercise. 30 minutes of aerobic exercise is recommended for at least 3 days per week to contribute to the regulation of both body composition, mood and to improve physical symptoms. Evidence suggests that it can be helpful in reducing symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 1-suffering from PMS (as determined by PMS scale) 2-Their ages range from 20 to 35 years 3-Having regular menstrual cycle

Exclusion Criteria:

* 1-Smoking 2-Following any special diet 3-Taking any medication 4-History of chronic disease 5-Having any psychiatric or gynecological problems

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: females with PMS will participate in this study with ages ranging from 20 to 35 years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Assessment of premenstrual syndrome | 5 minutes
  premenstrual syndrome scale consist of 2 sections and 19 questions about symptoms of PMS, it will be rated on the scale as not at all, mild, moderate or severe

SECONDARY OUTCOMES:
aerobic test | 6 minutes
  subject walk back and forth 6 times with maximum speed a distance of 35 meters, between every 35 meters, 10 seconds of rest will be considered

CONTACTS AND LOCATIONS:
Locations (1):
- Nisreen Ashraf, Giza, Egypt

REFERENCES:
- [Background] Hofmeister S, Bodden S. Premenstrual Syndrome and Premenstrual Dysphoric Disorder. Am Fam Physician. 2016 Aug 1;94(3):236-40. PMID 27479626
- [Background] Biggs WS, Demuth RH. Premenstrual syndrome and premenstrual dysphoric disorder. Am Fam Physician. 2011 Oct 15;84(8):918-24. PMID 22010771
- See also: premenstrual syndrome — https://pubmed.ncbi.nlm.nih.gov/12725453/